CLINICAL TRIAL: NCT06182124
Title: A Phase 1/2, Randomized, Double-Blind Trial of the Safety and Immunogenicity of a Multivalent Pneumococcal Conjugate Vaccine in Adults 18 Years of Age and Older
Brief Title: A Study to Learn About the Safety and Immune Response of a New Pneumococcal Vaccine in Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C4931001; NCT06182124 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-12-08; First posted 2023-12-26 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 (Stage 1): Multivalent Pneumococcal Vaccine - Formulation 1 (Experimental): Participants to receive a single injection of Multivalent Pneumococcal Vaccine - Formulation 1. This is a possible candidate for continuation in Phase 2 (Stage 2, 3, and 4).
  Interventions: Biological: Multivalent Pneumococcal Vaccine - Formulation 1
- Phase 1 (Stage 1): Multivalent Pneumococcal Vaccine - Formulation 2 (Experimental): Participants to receive a single injection of Multivalent Pneumococcal Vaccine - Formulation 2. This is a possible candidate for continuation in Phase 2 (Stage 2, 3, and 4).
  Interventions: Biological: Multivalent Pneumococcal Vaccine - Formulation 2
- Phase 1 (Stage 1) and Phase 2 (Stage 2): 20-valent pneumococcal conjugate vaccine (20vPnC) (Active Comparator): Participants to receive a single injection of 20vPnC.
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine (20vPnC)
- Phase 2 (Stage 3): a licensed pneumococcal comparator vaccine (Active Comparator): Participants to receive a single injection of a licensed pneumococcal comparator vaccine.
  Interventions: Biological: Licensed pneumococcal comparator vaccine
- Phase 2 (Stage 4): Multivalent Pneumococcal Vaccine - Formulation 3 (Experimental): Participants to receive a single injection of Multivalent Pneumococcal Vaccine - Formulation 3.
  Interventions: Biological: Multivalent Pneumococcal Vaccine - Formulation 3
- Phase 2 (Stage 4): Multivalent Pneumococcal Vaccine - Formulation 4 (Experimental): Participants to receive a single injection of Multivalent Pneumococcal Vaccine - Formulation 4.
  Interventions: Biological: Multivalent Pneumococcal Vaccine - Formulation 4

INTERVENTIONS:
Biological: Multivalent Pneumococcal Vaccine - Formulation 1 — Multivalent pneumococcal conjugate vaccine. This is a possible candidate for continuation in Phase 2 (Stages 2, 3, and 4).
  Arms: Phase 1 (Stage 1): Multivalent Pneumococcal Vaccine - Formulation 1
Biological: Multivalent Pneumococcal Vaccine - Formulation 2 — Multivalent pneumococcal conjugate vaccine. This is a possible candidate for continuation in Phase 2 (Stages 2, 3, and 4).
  Arms: Phase 1 (Stage 1): Multivalent Pneumococcal Vaccine - Formulation 2
Biological: 20-valent pneumococcal conjugate vaccine (20vPnC) — 20-valent pneumococcal conjugate vaccine (20vPnC)
  Other Names: Prevnar 20
  Arms: Phase 1 (Stage 1) and Phase 2 (Stage 2): 20-valent pneumococcal conjugate vaccine (20vPnC)
Biological: Licensed pneumococcal comparator vaccine — A licensed pneumococcal comparator vaccine
  Arms: Phase 2 (Stage 3): a licensed pneumococcal comparator vaccine
Biological: Multivalent Pneumococcal Vaccine - Formulation 3 — Multivalent pneumococcal conjugate vaccine
  Arms: Phase 2 (Stage 4): Multivalent Pneumococcal Vaccine - Formulation 3
Biological: Multivalent Pneumococcal Vaccine - Formulation 4 — Multivalent pneumococcal conjugate vaccine
  Arms: Phase 2 (Stage 4): Multivalent Pneumococcal Vaccine - Formulation 4

SUMMARY:
The purpose of this study is to learn about the safety and immune effects of a pneumococcal vaccine in adults. This vaccine can possibly provide protection against further pneumococcal disease.

This study will happen in 4 stages: Stage 1 is seeking participants who are between 18 years to 49 years of age. The participants will receive 1 of 2 pneumococcal vaccine candidates (different formulations) or 20vPnC (Prevnar 20) as a single shot given into the upper arm muscle.

Stage 2 will begin after participants have completed Stage 1, and a pneumococcal vaccine candidate has been decided.

Stage 2 is seeking participants who are adults 50 years of age and older. The participants will receive the chosen pneumococcal vaccine candidate from Stage 1 or 20vPnC (Prevnar 20). The vaccines will be given as a single shot into the upper arm muscle.

Stage 3 is seeking participants who are adults 50 years of age and older. The participants will receive the chosen pneumococcal vaccine candidate from Stage 1 or a licensed pneumococcal comparator vaccine. The vaccines will be given as a single shot into the upper arm muscle.

Stage 4 is seeking participants who are adults 50 years of age and older. The participants will receive either one of three pneumococcal vaccine candidates or one of two licensed pneumococcal comparator vaccines. The vaccines will be given as a single shot into the upper arm muscle.

Participants will take part in this study for about 6 months for Stage 1, Stage 3, and Stage 4 and 12 months for Stage 2. During this time participants will have from 2 to 4 clinic visits and 1 phone visit. At these clinic visits, participants will be asked if any side effects were experienced. The participants will also have to give blood samples during these clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥18 to<50 years of age (Stage 1) and ≥50 years of age (Stage 2, Stage 3, and Stage 4) at the time of consent
* Adults determined by clinical assessment to be eligible for the study, including adults with preexisting stable disease within 12 weeks before receipt of study intervention
* Participants willing to use acceptable contraception for at least 28 days after study intervention; female participants not of childbearing potential; male participants unable to father children
* Phase 1 (Stage 1): Adults 18 through 49 years of age with no history of ever receiving a pneumococcal vaccine (ie, pneumococcal vaccine-naïve)
* Phase 2 (Stages 2, 3, and 4): Adults ≥50 through 64 years of age with no history of ever receiving a pneumococcal vaccine (ie, pneumococcal vaccine-naïve) and adults 65 years of age and older with either no history of ever receiving a pneumococcal vaccine or who received PPSV23 >5 years prior to the first vaccination in this study (ie, experienced)

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction to any component in pneumococcal conjugate vaccines and any other diphtheria toxoid-containing vaccine
* Serious chronic disorder that in the investigator's opinion would make the participant inappropriate for entry into the study
* Medical or psychiatric condition (recent or active suicidal ideation/behavior or laboratory abnormality) that may increase risk of study participation or make participant inappropriate for the study
* Known or suspected immunodeficiency or other conditions associated with immunosuppression
* Planned receipt of any licensed or investigational pneumococcal vaccine, or planned receipt of any licensed or investigational pneumococcal vaccine through study participation
* Receipt of any inactivated or otherwise nonlive vaccine within 14 days or any live vaccine within 28 days before administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-05-23 (Estimated); Study Completion 2026-05-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prespecified local reactions within 7 days after vaccination | 7 days
  Prespecified local reactions (redness, swelling, and pain at the injection site) after vaccination
Percentage of participants reporting prespecified systemic events within 7 days after vaccination | 7 days
  Prespecified systemic events (fever, headache, fatigue, muscle pain, and joint pain) after vaccination
Percentage of participants reporting Adverse Events (AEs) within 1 month after vaccination | 1 month
  Adverse events occurring within 1 month after vaccination
Percentage of participants reporting Serious Adverse Events (SAEs) within 6 months after vaccination | 6 months
  SAEs occurring within 6 months after vaccination
Phase 2 (Stage 2) Only: Percentage of participants reporting related Serious Adverse Events (SAEs) through 12 months after vaccination | 12 months
  Related SAEs occurring through 12 months after vaccination

SECONDARY OUTCOMES:
Phase 1 (Stage 1) and Phase 2 (Stage 2) Only: Pneumococcal opsonophagocytic activity (OPA) geometric mean titers (GMTs) | 1 month after vaccination
  Pneumococcal OPA GMTs 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - Alliance for Multispecialty Research, LLC, Doral, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Optimal Research, Peoria, Illinois
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Headlands Research - Detroit, Southfield, Michigan
  - Rochester Clinical Research, LLC, Rochester, New York
  - Accellacare - Wilmington, Wilmington, North Carolina
  - AMR Clinical, Knoxville, Tennessee
  - Headlands Horizons LLC, Brownsville, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas
  - IMA Clinical Research San Antonio, San Antonio, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Sugar Land, Texas
  - DM Clinical Research, Tomball, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4931001